CLINICAL TRIAL: NCT04286958
Title: A Study of Camrelizumab As Consolidation Therapy After Radical Concurrent Chemoradiotherapy In Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Camrelizumab As Consolidation Therapy After Radical Concurrent Chemoradiotherapy In Locally Advanced ESCC
Acronym: ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Jun wang, Director, Hebei Medical University Fourth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRHB-CE001
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab (Experimental): All patients who had received radical concurrent chemoradiotherapy were treated with camrelizumab.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab: 200 mg was given intravenously over a period of 30 minutes (no less than 20 minutes and no longer than 60 minutes)

SUMMARY:
The purpose of this study is to assess efficacy and safety of patients who receive camrelizumab as consolidation therapy after radical concurrent chemoradiotherapy in locally advanced ESCC.

DETAILED DESCRIPTION:
In this study, 40 patients with locally advanced ESCC will be enrolled. All patients who had received radical concurrent chemoradiotherapy were treated with camrelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 75 years old;
2. Histology confirmed as esophageal squamous cell carcinoma;
3. T1bN+M0, T2-4N0-2M0 local progress period;
4. Have previously received radical concurrent chemoradiotherapy;
5. According to RECIST 1.1, at least one measurable lesion;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
7. Expected survival period ≥ 12 weeks;
8. Major organ function has to meet the following certeria:

1)For results of blood routine test HB≥90g/L; ANC≥1.5×109/L; PLT≥80×109/L; 2)For results of blood biochemical test ALB≥30g/L; ALT and AST<2.5×ULN; TBIL≤1.5ULN; Serum creatinine ≤1.5ULN; 9. Left ventricular ejection fraction (LVEF) ≥50%; 10. Women of childbearing age must have contraceptive measures or have test pregnancy (serum or urine) enroll the study before 14 days, and the results must be negative, and take the methods of contraception during the test and the last to have drugs after 8 weeks. Men must be contraception or has sterilization surgery during the test and the last to have drugs after 8 weeks; 11. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Subjects with immunosuppressive medications within 14 days of first administration of study treatment, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroid hormones (no more than 10 mg / day of prednisolone or other corticosteroids of equivalent pharmaceutical physiological dose);
2. The patient has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, Hyperthyroidism; patients with vitiligo; Asthma has been completely relieved in childhood, and patients who do not need any intervention after adulthood can be included; asthma patients who require bronchodilators for medical intervention cannot be included);
3. Patients with other malignant tumors within 5 years (except for the treated skin basal cell carcinoma and cervical carcinoma in situ);
4. Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV-DNA ≥1000 IU/ml) or hepatitis C (positive hepatitis C antibody, and HCV-RNA is higher than the lower limit of detection of the analytical method) or co-infection with hepatitis B and C, requiring antiviral treatment during the study ; 5.6 months before study drug administration, the following occurred: myocardial infarction, severe / unstable angina pectoris, grade III-IV cardiac insufficiency according to New York Heart Association(NYHA) criteria, uncontrolled arrhythmias (including QTcF interval male> 450 ms, female> 470 ms ,The QTcF interval is calculated using Fridericia formula), symptomatic congestive heart failure, cerebrovascular accidents (including transient ischemic attack or symptomatic pulmonary embolism);

6.Severe infections within 4 weeks before study drug administration (eg. Need intravenous drip antibiotics, antifungals or antivirals) or Unexplained fever>38.5℃ during screening visits or on the first scheduled day of dosing; 7.History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation; 8.Less than 4 weeks from the last clinical trial; 9.History of psychiatric drugs abuse and can't quit or patients with mental disorders; 10.The researchers think inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-12-22 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | evaluated in 24 months since the treatment began
  Baseline to measured date of progression or death from any cause

SECONDARY OUTCOMES:
Objective response rate (ORR) | tumor assessment every 6 weeks since the treatment began，up to 24 months
  Baseline to measured stable disease
Durarion of response (DOR) | tumor assessment every 6 weeks since the treatment began，up to 24 months
  From the first assessment to CR or PR to the first assessment to PD or death from any cause
Overall survival (OS) | the first day of treatment to death or last survival confirm date,up to 24 months
  Baseline to measured date of death from any cause
Adverse events | up to 24 months
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03. The number of Participants with adverse events will be recorded at each treatment visit

OTHER OUTCOMES:
Biomarkers | up to 24 months
  Relationship between tumor markers and efficacy in tumor tissues and peripheral blood (including but not limited to PD-L1, TMB, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China